CLINICAL TRIAL: NCT03627130
Title: Effect of Inorganic Nitrate on Contrast-induced Nephropathy in Patients Undergoing Coronary Angiography/Percutaneous Coronary Intervention for Acute Coronary Syndrome (ACS): A Randomised Single-centre, Double-blind Placebo-controlled Trial
Brief Title: The Use of Inorganic Nitrate for the Prevention of Contrast-induced Nephropathy
Acronym: NITRATE-CIN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Barts & The London NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 18/1
Record Dates: First submitted 2018-01-17; First posted 2018-08-13 (Actual); Last update posted 2022-12-16 (Actual); Status verified 2022-12

CONDITIONS: Contrast-induced Nephropathy; Acute Kidney Injury; Acute Coronary Syndrome
Keywords: Percutaneous Coronary Intervention; Nitric Oxide; Nitrite; Acute Kidney Injury; Acute Coronary Syndrome
MeSH Terms: conditions — Acute Kidney Injury; Acute Coronary Syndrome | interventions — potassium nitrate; Potassium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: IMP and placebo will be identical
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Potassium Nitrate (Active Comparator): Potassium nitrate capsules (KNO3: 12 mmol giving 744 mg of nitrate) for 5 days
  Interventions: Drug: Potassium Nitrate
- Potassium Chloride (Placebo Comparator): Potassium Chloride
  Interventions: Drug: Potassium Chloride

INTERVENTIONS:
Drug: Potassium Nitrate — Potassium nitrate capsules (KNO3: 12 mmol giving 744 mg of nitrate) for 5 days
  Arms: Potassium Nitrate
Drug: Potassium Chloride — Potassium Chloride capsules for 5 days
  Arms: Potassium Chloride

SUMMARY:
Contrast-induced nephropathy (CIN), an acute kidney injury resulting from the administration of intravascular iodinated contrast media, is an important cause of morbidity/mortality following coronary angiographic procedures in high-risk patients. Despite preventative measures intended to mitigate the risk of CIN, there remains a need for an effective intervention. Dietary inorganic nitrate therapy, which through its chemical reduction in the body delivers nitric oxide has shown promise in attenuating CIN, but its effectiveness in preserving long-term renal function is unknown.

DETAILED DESCRIPTION:
The NITRATE-CIN trial is a single-centre, randomised double-blinded placebo-controlled trial, which plans to recruit, over a period of 2 years, 640 patients presenting with acute coronary syndromes (ACS) who are at risk of CIN.

Patients will be randomised to either dietary inorganic nitrate therapy or placebo.

The primary endpoint will be the development of CIN (KDIGO criteria). A key secondary endpoint will be whether nitrate therapy impacts upon persistent renal impairment over a 3-month follow-up period. Additional secondary endpoints include the measurement of serum renal biomarkers (e.g. neutrophil gelatinase-associated lipocalin) and urinary albumin at 6, 48 h and 3 months following administration of contrast.

Findings from NITRATE-CIN will potentially demonstrate that nitrate attenuates contrast-induced acute and chronic kidney injury and influence future clinical practice guidelines in at-risk patients undergoing coronary angiographic procedures.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing coronary angiography+/-Percutaneous Coronary Intervention (PCI) for NSTE-ACS
2. Requirement for CIN prophylaxis as per Barts Heart Centre Criteria for CIN prophylaxis:

   eGFR<60ml/min OR 2 of the following: diabetes, liver failure (cirrhosis), age > 70yr, exposure to contrast in last 7 days, heart failure (or LVEF<40%), concomitant renally active drugs (ACEi, ARB, NSAIDs, aminoglycosides, diuretics)
3. Aged >18
4. Patients able and willing to give their written informed consent.

Exclusion Criteria:

1. ST segment myocardial infarction undergoing Primary PCI.
2. Patients with eGFR<30ml/min or on renal replacement therapy
3. Subjects presenting with cardiogenic shock (systolic blood pressure <80 mmHg for >30 minutes, or requiring inotropes or emergency intra aortic balloon pump for hypotension treatment) or cardiopulmonary resuscitation
4. Current life-threatening condition other than vascular disease that may prevent a subject completing the study.
5. Use of an investigational device or investigational drug within 30 days or 5 half-lives (whichever is the longer) preceding the first dose of study medication.
6. Patients considered unsuitable to participate by the research team (e.g., due to medical reasons, laboratory abnormalities, or subject's unwillingness to comply with all study related procedures).
7. Severe acute infection
8. Pregnancy
9. Breast-feeding mothers.
10. Any Inclusion Criteria not met

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 640 (Actual)
Dates: Start 2018-11-29 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2022-05-30 (Actual)

PRIMARY OUTCOMES:
Contrast Induced Nephropathy | 48-72 hours
  Defined by Kidney Disease: Improving Global Outcomes (KDIGO) criteria

SECONDARY OUTCOMES:
Demonstration of a persistent benefit of dietary inorganic nitrate against long-term renal impairment | 3 months
  Difference in real function as measured by eGFR (estimated glomerular filtration rate) at 3 months post-contrast exposure
Measurement of Circulating Nitrite and Nitrate levels | Baseline, and at 6 hours, 48 hours and 3 months following treatment.
  Plasma Nitrite/Nitrate levels
Major Adverse Cardiac Events | 3 and 12 months follow-up
  Defined as death, non-fatal myocardial infarction, revascularisation, acute heart failure, non-fatal stroke
Cost effectiveness of dietary inorganic Nitrate | 1 year
  Incremental Cost Effectiveness Ratio (ICER)
To determine if dietary inorganic nitrate ingestion decreases sub-clinical renal injury as measured by urinary renal biomarkers | 4-6 hours
  Measurement of urinary IGFB7/TIMP-2
To determine if dietary inorganic nitrate ingestion decreases sub-clinical renal injury as measured by serum biomarkers | 4-6 hours
  Measurement of serum Neutrophil gelatinase-associated lipocalin (NGAL)
To determine if dietary inorganic nitrate decreases rates of post-procedural Myocardial Infarction | 6-12 hrs
  Definition as per Society for Cardiovascular Angiography and Interventions (SCAI)

CONTACTS AND LOCATIONS:
Overall Officials: Amrita Ahluwalia, PhD, Principal Investigator — Queen Mary University of London
Locations (1):
- Barts Heart Centre, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
The trial protocol will be published prior to the commencement of the study
Supporting Information: Study Protocol
Time Frame: Mid-late 2018
Access Criteria: Freely available via journal

REFERENCES:
- [Derived] Jones DA, Beirne AM, Kelham M, Wynne L, Andiapen M, Rathod KS, Parakaw T, Adams J, Learoyd A, Khan K, Godec T, Wright P, Antoniou S, Wragg A, Yaqoob M, Mathur A, Ahluwalia A. Inorganic nitrate benefits contrast-induced nephropathy after coronary angiography for acute coronary syndromes: the NITRATE-CIN trial. Eur Heart J. 2024 May 13;45(18):1647-1658. doi: 10.1093/eurheartj/ehae100. PMID 38513060
- [Derived] Beirne AM, Mitchelmore O, Palma S, Andiapen M, Rathod KS, Hammond V, Bellin A, Cooper J, Wright P, Antoniou S, Yaqoob MM, Naci H, Mathur A, Ahluwalia A, Jones DA. NITRATE-CIN Study: Protocol of a Randomized (1:1) Single-Center, UK, Double-Blind Placebo-Controlled Trial Testing the Effect of Inorganic Nitrate on Contrast-Induced Nephropathy in Patients Undergoing Coronary Angiography for Acute Coronary Syndromes. J Cardiovasc Pharmacol Ther. 2021 Jul;26(4):303-309. doi: 10.1177/1074248421000520. Epub 2021 Mar 25. PMID 33764198